CLINICAL TRIAL: NCT03351153
Title: Prediction of the Collapse of Necrotic Femoral Head Using Computed Tomography Scan and X-ray Before Hip Arthroplasty: Study Protocol for a Single-center, Open-label, Diagnostic Trial
Brief Title: Prediction of the Collapse of Necrotic Femoral Head Using Computed Tomography Scan and X-ray Before Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Principal Investigator, Di Qin, Principal Investigator, Hebei Medical University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HebeiMUth-001
Record Dates: First submitted 2017-11-13; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Hip Arthropathy
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- X-ray group (Other): In the X-ray group, the changes in femoral head height were measured with X-ray in an anteroposterior position of the pelvis (healthy and affected sides of the hip) at preoperative 1 week.
  Interventions: Radiation: X-ray
- CT group (Other): In the CT group, changes of femoral head height were measured with CT scan on bilateral hips (healthy side and affected side) at preoperative 1 week.
  Interventions: Radiation: CT
- Specimen group (Other): In the specimen group, femoral head on the affected side was resected during surgery and directly measured with a ruler and vernier caliper.
  Interventions: Other: specimen

INTERVENTIONS:
Radiation: X-ray — In the X-ray group, the changes in femoral head height were measured with X-ray in an anteroposterior position of the pelvis (healthy and affected sides of the hip) at preoperative 1 week
  Arms: X-ray group
Radiation: CT — In the CT group, changes of femoral head height were measured with CT scan on bilateral hips (healthy side and affected side) at preoperative 1 week
  Arms: CT group
Other: specimen — In the specimen group, femoral head on the affected side was resected during surgery and directly measured with a ruler and vernier caliper.
  Arms: Specimen group

SUMMARY:
To verify that CT scan and X-ray can predict the collapse of the necrotic femoral head before hip arthroplasty and effectively guide the surgical management.

DETAILED DESCRIPTION:
Osteonecrosis of the femoral head (ONFH) is a common and frequently occurring disease. The main clinical manifestations are hip pain and dysfunction. The etiology and pathogenesis of ONFH caused by various reasons are the problems that have not been solved yet in the field of orthopedics. If want to achieve satisfactory therapeutic effect, surgical choice is essential. It is very important for prognosis to master the indications of operation and take appropriate treatment measures, especially the great difference between palliative surgery and hip arthroplasty.

To determine whether the femoral head collapses and the degree of collapse of the articular cartilage of the femoral head can help physicians to select an optimal surgical plan. Chinese scholars commonly believe that if the femoral head collapse is less than 2 mm, investigators can choose autologous bone graft, allogeneic bone graft and other palliative surgery. If the femoral head collapse is more than 2 mm, investigators can choose total hip arthroplasty. However, above standard has not been extensively accepted worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ONFH confirmed preoperatively (FICAT stages III and IV; Appendix 1)14
* Unilateral total hip arthroplasty
* Age range: 32-68 years
* Irrespective of sex
* Sign the informed consent

Exclusion Criteria:

* Infection
* Tuberculosis
* Tumor
* Severe osteoporosis

Ages: 32 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-07-08 (Actual); Primary Completion 2012-01-04 (Actual); Study Completion 2012-01-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity | At preoperative 1 week
  Sensitivity refers to true positive rate, the percentage of patients with actual illness who was correctly diagnosed in overall patients. High sensitivity indicated high correct rate of femoral head collapse.

SECONDARY OUTCOMES:
Specificity | At preoperative 1 week
  Specificity refers to true negative rate, the percentage of patients with actual disease-free who are correctly judged as disease-free according to the diagnostic criteria. The high specificity indicates high accuracy of diagnosis.
positive predictive value | At preoperative 1 week
  Positive predictive value refers to the proportion of patients with actual illness among all positive cases, can reflect the possibility of affecting target disease in patients with positive screening test result.
Negative predictive value | At preoperative 1 week
  Negative predictive value refers to the proportion of patients with negative screening test result who do not suffer from diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Di Qin, Principal Investigator — Third Hospital of Hebei Medical University